CLINICAL TRIAL: NCT05945927
Title: An Observational Study to Evaluate the Safety and Effectiveness of Trastuzumab Emtansine (T-DM1) as Second- or Later-Line Therapy in Chinese Patients With HER2 Positive Advanced Breast Cancer
Brief Title: A Study to Evaluate the Safety and Effectiveness of Trastuzumab Emtansine (T-DM1) as Therapy in Chinese Participants With HER2 Positive Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML44675
Record Dates: First submitted 2023-06-29; First posted 2023-07-14 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with HER2-positive Advanced Breast Cancer: Participants will be prospectively followed from the index date (the first treatment of T-DM1) for up to 1 year.
  Interventions: Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Trastuzumab emtansine — Trastuzumab emtansine will be administered as per local clinical practice and local labeling.
  Other Names: T-DM1

SUMMARY:
This study is a post-marketing, observational, multicenter, prospective study. It will investigate the the safety and effectiveness of T-DM1 in the Chinese population in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HER2-positive, unresectable locally advanced or metastatic breast cancer before the start of T-DM1 treatment
* Had prior treatment for breast cancer which must contain a taxane and trastuzumab
* Get the treatment of T-DM1 for the first time after diagnosis of breast cancer

Exclusion Criteria:

* Patients not receiving treatment for HER2-positive breast cancer with T-DM1 according to standard of care and in line with the current summary of product characteristics (SPC)/local labeling
* Has been previously treated with T-DM1 before current clinical visit
* Currently participating in any clinical trials
* Previously participated in any clinical trials investigating anti-HER2 drug within 1 year of the initiation of T-DM1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of HER2-positive advanced breast cancer will be included in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Up to approximately 1 year from index date

SECONDARY OUTCOMES:
Real-world Progression Free Survival (rwPFS) | From the index date to the date of first progression of disease as recorded in rwTR or death due to any reason, whichever occurs first (up to approximately 1 year from index date)
Time-to-treatment Discontinuation (TTD) | Up to approximately 1 year from index date
Percentage of Participants Exposed to T-DM1 by Line of Therapy | Up to approximately 1 year from index date
Percentage of Participants Exposed to T-DM1 by Dosage | Up to approximately 1 year from index date
Percentage of Participants Exposed to T-DM1 by Dose Intensity | Up to approximately 1 year from index date
Percentage of Participants Exposed to T-DM1 by Duration | Up to approximately 1 year from index date
Percentage of Participants Exposed to Prior and Concomitant Medication by WHODrug Anatomical Therapeutic Chemical (ATC) Classification System | Up to approximately 1 year from index date
Percentage of Participants Exposed to Prior and Concomitant Surgery/Procedure by Medical Dictionary for Regulatory Activities (MedDRA) | Up to approximately 1 year from index date

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- China (30):
  - Anyang Tumor Hosptial, Anyang
  - Affiliated Hospital of Hebei University, Baoding
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Beijing Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Province Cancer Hospital, Hefei
  - Jiangmen Central Hospital, Jiangmen
  - The First Affiliated Hospital Of Shandong First Medical University, Jinan
  - Dongyang People's Hospital, Jinhua
  - The Third Hospital of Nanchang, Nanchang
  - Nanjing Gulou Hospital, Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Affiliated Hospital of Nantong University, Nantong
  - Ningbo No.2 Hospital, Ningbo
  - China Medical University (CMU) First Affiliated Hospital, Shenyang
  - Cancer Hospital Chinese Academy of Medical Sciences Shenzhen Center, Shenzhen
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Tianjin Cancer Hospital, Tianjin
  - Cancer Hospital Affliated to Xinjiang Medical University, Ürümqi
  - Weifang People's Hospital, Weifang
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Yibin Second People's Hospital, Yibin
  - Zhejiang Cancer Hospital, Zhejiang

IPD SHARING:
Plan to Share IPD: No